CLINICAL TRIAL: NCT02616029
Title: A Phase 3b Open-Label Pilot Study to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Fixed Dose Combination (FDC) in Virologically-Suppressed HIV-1 Infected Adult Subjects Harboring the Archived Isolated NRTI Resistance Mutation M184V/M184I
Brief Title: Study to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Fixed Dose Combination (FDC) in Virologically-Suppressed HIV-1 Infected Adults Harboring the Archived Isolated NRTI Resistance Mutation M184V/M184I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1824; 2015-002710-74 (EudraCT Number)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: E/C/F/TAF (Experimental): Participants with M184V and/or M184I mutations in reverse transcriptase and without any other NRTI resistance mutation switched from their current human immunodeficiency virus (HIV) treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
  Allowed third agents include: lopinavir/ritonavir (LPV/r), atazanavir + ritonavir (ATV+RTV), atazanavir+cobicistat (ATV+COBI), darunavir + ritonavir (DRV+RTV), darunavir + cobicistat (DRV+COBI), fosamprenavir + ritonavir (FPV + RTV), saquinavir + ritonavir (SQV + RTV), atazanavir (ATV) (no booster) efavirenz (EFV), rilpivirine (RPV), nevirapine (NVP), etravirine (ETR), raltegravir (RAL) or dolutegravir (DTG).
  Interventions: Drug: E/C/F/TAF
- Part 2: E/C/F/TAF (Experimental): Participants with M184V and/or M184I mutations in reverse transcriptase and with or without 1 or 2 TAMs switched from their current HIV treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
  Allowed third agents include: LPV/r, ATV+RTV, ATV+COBI, DRV+RTV, DRV+COBI, FPV + RTV, SQV + RTV, ATV (no booster) EFV, RPV, NVP, ETR, RAL or DTG.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablets administered orally once daily
  Other Names: Genvoya®

SUMMARY:
The primary objective of the study is to evaluate the efficacy of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) after switching from a stable regimen consisting of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) or abacavir/lamivudine (ABC/3TC) plus a third antiretroviral (ARV) agent in participants harboring the archived nucleoside/nucleotide reverse transcriptase inhibitor (NRTI) resistance mutation M184V and/or M184I in human immunodeficiency virus (HIV) -1 reverse transcriptase.

This is a two part study. If the rate of virologic failure in Part 1 is deemed acceptable, once the internal data monitoring committee officially completes the interim review, the study will continue to Part 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented historical genotype report showing mutation M184V and/or M184I (mixtures are acceptable) in reverse transcriptase. Individuals must not have any primary integrase strand transfer inhibitor (INSTI) or primary protease inhibitor (PI) resistance mutations present on historical genotype; non-nucleoside reverse transcriptase inhibitor (NNRTI) mutations are allowed.
* Proviral deoxyribonucleic acid (DNA) test must not have additional exclusion resistance mutations against PIs, NRTIs and INSTIs

  * Part 1: Historical genotype report must show mutation M184V and/or M184I in reverse transcriptase WITHOUT any other NRTI resistance mutation (including thymidine analogue-associated mutations [TAMs] [TAMs are: M41L, D67N, K70R, L210W, T215Y/F, and K219Q/E/N/R], K65R, K70E, T69 insertion, and Q151M mutation complex [A62V, V75I, F77L, F116Y, Q151M])
  * Part 2 (after the interim efficacy review): Historical genotype report must show M184V and/or M184I in reverse transcriptase WITH or WITHOUT 1 or 2 TAMs. Evidence of K65R, K70E, T69 insertion and/or Q151M mutation complex will not be eligible
* Currently receiving an ARV regimen consisting of FTC/TDF or ABC/3TC in combination with one third ARV agent for ≥ 6 consecutive months preceding the screening visit
* Documented plasma HIV-1 ribonucleic acid (RNA) levels < 50 copies/mL for ≥ 6 months preceding the screening visit
* Plasma HIV-1 RNA levels < 50 copies/mL at screening visit
* Estimated glomerular filtration rate (GFR) ≥ 30 mL/min according to the Cockcroft-Gault formula for creatinine clearance
* A female individual is eligible to enter the study if it is confirmed that she is:

  * not pregnant
  * of non-childbearing potential
  * stopped menstruating for ≥ 12 months
  * of childbearing potential and agrees to utilize the protocol-specified method of contraception or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following discontinuation of study drugs
* Male individuals must agree to use the protocol-specified method(s) of contraception during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from screening throughout the study period and for 30 days following the last study drug dose

  * Male individuals must agree to refrain from sperm donation from first dose until at least 30 days after the last study drug dose

Key Exclusion Criteria:

* Individuals will have no evidence of previous virologic failure on a PI/r or INSTI-based regimen (with or without resistance to either class of ARV). Individuals may have evidence of prior virologic failure on only an NNRTI plus 2 NRTI-based regimen
* Individuals on a current PI/r-based regimen will have no evidence of previous use of any approved or experimental integrase strand transfer inhibitor (INSTI) (for any length of time)
* Hepatitis C infection that would require therapy during the study
* Hepatitis B surface antigen (HBsAg) positive
* Individuals with clinical evidence of decompensated cirrhosis (eg, ascites, encephalopathy, variceal bleeding)
* Have an implanted defibrillator or pacemaker
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non invasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Day 1 and must not be anticipated to require systemic therapy during the study
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (3):
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
- France (7):
  - Hopital Sainte Marguerite - Hospital, Marseille
  - CHU de Nantes, Nantes
  - CHU de Nice-l Archet, Nice
  - CHR Orleans la Source, Orléans
  - Hopital Saint Louis, Paris
  - Hopital Necker les Enfants Malades, Paris
  - CHU Tours Service de Médecine Internes et Maladies Infectieuses, Tours
- Germany (3):
  - Universitatsklinikum Essen, Essen
  - ICH Study Center- Dedicated Research, Hamburg
  - Universitat Mainz, Mainz
- Italy (4):
  - IRCCS A.O.U. San Martino, Genova
  - Fondazione IRCCS San Raffaele del Monte Tabor, Milan
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan
  - Comprensorio Amedeo Di Savoia Birago Di Vische, Torino
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona - Hospital, Barcelona
  - Hospital Universitario 12 de Octubre - Hospital, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Perez-Valero I, Llibre JM, Lazzarin A, di Perri G, Pulido F, Molina JM, Esser S, Margot N, Shao Y, Piontkowsky D, Das M, McNicholl IR, Haubrich R. A Phase 3b Open-Label Pilot Study to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) in Virologically-Suppressed HIV-1 Infected Adults Harboring the NRTI Resistance Mutation M184V/I (GS-US-292-1824): Week 24 Results [Poster PE13/20]. 17th European AIDS Conference (EACS), 6-9 November 2019, Basel, Switzerland.
- [Background] Perez-Valero I, Llibre JM, Lazzarin A, di Perri G, Pulido F, Molina JM, Esser S, McNicholl IR, Lorgeoux RP, Margot N, Shao Y, Piontkowsky D, Das M, Haubrich R. A Phase 3b Open-Label Pilot Study to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Single-Tablet Regimen in Virologically-Suppressed HIV-1 Infected Adults Harboring the NRTI Resistance Mutation M184V and/or M184I (GS-US-292-1824): Week 24 Results [Oral abstract]. 22nd International AIDS Conference, 23-27 July 2018, Amsterdam, The Netherlands.
- [Background] Perez-Valero I, Llibre JM, Lazzarin A, di Perri G, Pulido F, Molina JM, Esser S, McNicholl IR, Lorgeoux RP, Margot N, Shao Y, Piontkowsky D, Das M, Haubrich R. A Phase 3b Open-Label Pilot Study to Evaluate Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Single Tablet Regimen in Virologically-Suppressed HIV-1 Infected Adults Harboring the NRTI Resistance Mutation M184V and/or M184I (GS-US-292-1824): Week 12 Results [Poster]. XXVI International Workshop on HIV Drug Resistance and Treatment Strategies, 6-8 November 2017, Johannesburg, South Africa.
- [Derived] Perez-Valero I, Llibre JM, Castagna A, Pulido F, Molina JM, Esser S, Margot N, Shao Y, Temme L, Piontkowsky D, McNicholl IR, Haubrich R. Switching to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide in Adults With HIV and M184V/I Mutation. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):490-495. doi: 10.1097/QAI.0000000000002595. PMID 33315694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Europe. The first participant was screened on 17 December 2015. The last study visit occurred on 11 July 2019.
Pre-assignment Details: 120 participants were screened.
Groups:
- Part 1: E/C/F/TAF: Participants with M184V and/or M184I mutations in reverse transcriptase and without any other nucleos(t)ide reverse transcriptase inhibitor (NRTI)-resistance mutation switched from their current human immunodeficiency virus (HIV) treatment regimen consisting of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) or abacavir/lamivudine (ABC/3TC) plus a third antiretroviral agent to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet orally once daily for 48 weeks.
- Part 2: E/C/F/TAF: Participants with M184V and/or M184I mutations in reverse transcriptase and with or without 1 or 2 thymidine analog-associated mutations (TAMs) switched from their current HIV treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
Period: Overall Study
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF
Started | 38 | 28
Completed | 34 | 26
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Not completed — Enrolled and Never Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Part 1: E/C/F/TAF: Participants with M184V and/or M184I mutations in reverse transcriptase and without any other NRTI-resistance mutation switched from their current human immunodeficiency virus (HIV) treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
- Part 2: E/C/F/TAF: Participants with M184V and/or M184I mutations in reverse transcriptase and with or without 1 or 2 TAMs switched from their current HIV treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total
Number analyzed (Participants) | 37 | 27 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9.2) | 52 (9.5) | 51 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 29 | 18 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For participants in Not Permitted category: local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 6 | 4 | 10
    Ethnicity: Not Hispanic or Latino | 27 | 21 | 48
    Ethnicity: Not Permitted | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For participants in Not Permitted category: local regulators did not allow collection of ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0
    Race: Asian | 0 | 0 | 0
    Race: Black | 7 | 8 | 15
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0
    Race: White | 27 | 17 | 44
    Race: Not Permitted | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8
  Italy | 2 | 3 | 5
  France | 14 | 15 | 29
  Germany | 4 | 1 | 5
  Spain | 14 | 3 | 17
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 1.29 (0.056) | 1.29 (0.046) | 1.29 (0.052)
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  < 50 copies/mL | 37 | 27 | 64
  ≥ 50 copies/mL | 0 | 0 | 0
Cluster Determinant 4+ (CD4+) Cell Count [Mean (Standard Deviation); unit: cells/µL] | 740 (319.6) | 665 (312.7) | 708 (316.4)
CD4+ Cell Count Categories [Count of Participants; unit: Participants]
  < 50 cells/µL | 0 | 0 | 0
  ≥ 50 to < 200 cells/µL | 1 | 2 | 3
  ≥ 200 to < 350 cells/µL | 3 | 1 | 4
  ≥ 350 to < 500 cells/µL | 4 | 5 | 9
  ≥ 500 cells/µL | 29 | 19 | 48
HIV Disease Status [Count of Participants; unit: Participants]
  Asymptomatic | 30 | 23 | 53
  Symptomatic HIV Infection | 4 | 1 | 5
  Acquired Immune Deficiency Syndrome (AIDS) | 3 | 3 | 6
CD4 Percentage (%) [Mean (Standard Deviation); unit: percentage of CD4 cells] | 32.9 (10.12) | 31.2 (11.43) | 32.2 (10.63)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) < 50 Copies/mL at Week 12 as Defined by Pure Virologic Response (PVR)
Description: The percentage of participants with PVR for HIV-1 RNA cutoff at 50 copies/mL at Week 12 was summarized. PVR was the percentage of participants who did not have a confirmed virologic rebound. Virologic rebound was defined as 2 consecutive HIV-1 RNA values ≥ 50 copies/mL or the last available HIV-1 RNA value ≥ 50 copies/mL during the study followed by premature discontinuation from the study.
Time Frame: Week 12
Population: The Full Analysis Set included all the randomized participants who received at least one dose of study drug and excluded participants with any major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: E/C/F/TAF: Participants with M184V and/or M184I mutations in reverse transcriptase and without any other NRTI-resistance mutation switched from their current HIV treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
- Total E/C/F/TAF: Participants switched from their current HIV treatment regimen consisting of FTC/TDF or ABC/3TC plus a third antiretroviral agent to E/C/F/TAF (150/150/200/10 mg) FDC tablet orally once daily for 48 weeks.
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 100.0 [90.3 to 100.0] | 100.0 [86.8 to 100.0] | 100.0 [94.2 to 100.0]

2. Secondary Outcome: Percentage of Participants With Emergence of New Mutations in HIV-1 Reverse Transcriptase and Integrase
Description: Development of new resistance mutations was assessed in participants who developed virologic failure, defined as 2 consecutive HIV-1 RNA result ≥ 50 copies/mL at any point in the study or with HIV-1 RNA ≥ 50 copies/mL at last visit.
Time Frame: Day 1 up to 48 weeks
Population: Participants in the Full Analysis Set were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 Using PVR
Description: The percentage of participants with PVR for HIV-1 RNA cutoff at 50 copies/mL at Week 24 was summarized. PVR was the percentage of participants who did not have a confirmed virologic rebound. Virologic rebound was defined as 2 consecutive HIV-1 RNA values ≥ 50 copies/mL or the last available HIV-1 RNA value ≥ 50 copies/mL during the study followed by premature discontinuation from the study.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 100.0 [90.3 to 100.0] | 100.0 [86.8 to 100.0] | 100.0 [94.2 to 100.0]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 Using PVR
Description: The percentage of participants with PVR for HIV-1 RNA cutoff at 50 copies/mL at Week 48 was summarized. PVR was the percentage of participants who did not have a confirmed virologic rebound. Virologic rebound was defined as 2 consecutive HIV-1 RNA values ≥ 50 copies/mL or the last available HIV-1 RNA value ≥ 50 copies/mL during the study followed by premature discontinuation from the study.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 100.0 [90.3 to 100.0] | 100.0 [86.8 to 100.0] | 100.0 [94.2 to 100.0]

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 12 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 12 window was between Day 71 and 98 (inclusive).
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 91.7 [77.5 to 98.2] | 96.2 [80.4 to 99.9] | 93.5 [84.3 to 98.2]

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 24 window was between Day 141 and 210 (inclusive).
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 91.7 [77.5 to 98.2] | 100.0 [86.8 to 100.0] | 95.2 [86.5 to 99.0]

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 12 window was between Day 295 and 378 (inclusive).
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 88.9 [73.9 to 96.9] | 96.2 [80.4 to 99.9] | 91.9 [82.2 to 97.3]

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 12 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 20 copies/mL at Week 12 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 12 window was between Day 71 and 98 (inclusive).
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 91.7 [77.5 to 98.2] | 96.2 [80.4 to 99.9] | 93.5 [84.3 to 98.2]

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 24 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 20 copies/mL at Week 24 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 24 window was between Day 141 and 210 (inclusive).
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 88.9 [73.9 to 96.9] | 100.0 [86.8 to 100.0] | 93.5 [84.3 to 98.2]

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 48 Using the FDA Snapshot Analysis
Description: The percentage of participants with HIV-1 RNA < 20 copies/mL at Week 48 was also analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 12 window was between Day 295 and 378 (inclusive).
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 88.9 [73.9 to 96.9] | 96.2 [80.4 to 99.9] | 91.9 [82.2 to 97.3]

11. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 Using the Missing = Failure (M = F) Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 12 was analyzed using the M = F approach. In this approach, all missing data was treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 97.2 [85.5 to 99.9] | 96.2 [80.4 to 99.9] | 96.8 [88.8 to 99.6]

12. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 Using the M = F Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the M = F approach. In this approach, all missing data was treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 91.7 [77.5 to 98.2] | 100.0 [86.8 to 100.0] | 95.2 [86.5 to 99.0]

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 Using the M = F Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the M = F approach. In this approach, all missing data was treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 36 | 26 | 62
percentage of participants | 91.7 [77.5 to 98.2] | 96.2 [80.4 to 99.9] | 93.5 [84.3 to 98.2]

14. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 Using the Missing = Excluded (M = E) Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 12 was also analyzed using the M = E approach. In this approach, all missing data was excluded in the computation of the proportions.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 35 | 26 | 61
percentage of participants | 100.0 [90.0 to 100.0] | 96.2 [80.4 to 99.9] | 98.4 [91.2 to 100.0]

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 Using the M = E Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was also analyzed using the M = E approach. In this approach, all missing data was excluded in the computation of the proportions.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 26 | 59
percentage of participants | 100.0 [89.4 to 100.0] | 100.0 [86.8 to 100.0] | 100.0 [93.9 to 100.0]

16. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 Using the M = E Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was also analyzed using the M = E approach. In this approach, all missing data was excluded in the computation of the proportions.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 25 | 58
percentage of participants | 100.0 [89.4 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [93.8 to 100.0]

17. Secondary Outcome: Change From Baseline in Cluster Determinant 4+ (CD4+) Cell Count at Week 12
Time Frame: Baseline (Day 1); Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 25 | 58
cells/µL | -47 (194.1) | -6 (116.1) | -30 (165.1)

18. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline (Day 1); Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 26 | 59
cells/µL | -40 (162.1) | 28 (212.5) | -10 (187.4)

19. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline (Day 1); Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 31 | 25 | 56
cells/µL | -6 (131.9) | 27 (120.4) | 9 (126.8)

20. Secondary Outcome: Change From Baseline in CD4 Percentage (%) at Week 12
Time Frame: Baseline (Day 1); Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 25 | 58
percentage of CD4 cells | -0.4 (3.37) | 1.5 (3.01) | 0.4 (3.33)

21. Secondary Outcome: Change From Baseline in CD4 % at Week 24
Time Frame: Baseline (Day 1); Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 33 | 26 | 59
percentage of CD4 cells | 0.1 (3.25) | 1.1 (4.30) | 0.5 (3.75)

22. Secondary Outcome: Change From Baseline in CD4 % at Week 48
Time Frame: Baseline (Day 1); Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Part 1: E/C/F/TAF | Part 2: E/C/F/TAF | Total E/C/F/TAF
Number analyzed (Participants) | 31 | 25 | 56
percentage of CD4 cells | 0.2 (3.12) | 1.5 (3.64) | 0.8 (3.39)

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum: 48 Weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug. Safety data for overall study population is presented in this section as all participants received same treatment.
Arm/Group | Total E/C/F/TAF
All-Cause Mortality (participants affected / at risk) | 1/64
Serious Adverse Events (participants affected / at risk) | 5/64
Other Adverse Events (participants affected / at risk) | 26/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total E/C/F/TAF (N=64)
Death (General disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total E/C/F/TAF (N=64)
Diarrhoea (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 7
Bronchitis (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT02616029/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT02616029/SAP_002.pdf